CLINICAL TRIAL: NCT03422224
Title: Alloreactive t Cell Repertoire in Kidney Transplantation Recipients
Brief Title: ALLoreactive T-Cell receptOr RePertoire in kidnEy tranSplantation
Acronym: ALL-T-COPIES
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Rainer Oberbauer, Prof. Dr, Medical University of Vienna
Other Study IDs: ALL-T-COPIES
Record Dates: First submitted 2018-01-30; First posted 2018-02-05 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Renal Transplant Rejection; Immune Repertoire; Transplant; Complication, Rejection; Alloreactivity
MeSH Terms: conditions — Rejection, Psychology | interventions — Lymphocyte Culture Test, Mixed

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — PBMC needle biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Good transplant function: Kidney transplant recipients without histological signs of rejection.
  Interventions: Diagnostic Test: Mixed lymphocyte reaction
- Transplant Rejection: Kidney transplant recipinets experiencing a T cell mediated rejection episode.
  Interventions: Diagnostic Test: Mixed lymphocyte reaction

INTERVENTIONS:
Diagnostic Test: Mixed lymphocyte reaction — Assessment of alloreactive T cell repertoire

SUMMARY:
In this study, the investigators will establish a workflow to generate unique patterns of the donor-reactive T cell repertoire using mixed lymphocyte reactions to select alloreactive T cell clones prior to transplantation Tissue infiltrating as well as blood bound T cells will be characterized based on:

1. Identification of donor-specific T cell receptor sequences pre- and post-transplant by in vitro expansion to determine unique patterns
2. Quantification and comparison of donor-specific T cell clones in kidney biopsy and blood samples.
3. Analysis of the TCR repertoire diversities derived from kidney biopsy and blood samples and association of repertoire diversities with the histomorphological phenotype of T cell mediated rejection.
4. Identification of T cell subtypes within the donor-reactive population. The investigators specifically hypothesize that highly expanded donor-reactive T cell clones in both kidney tissue and blood samples at time of indication biopsy are associated with the histological phenotype of acute T cell mediated rejection. The investigators have previously shown that there is a strong correlation between highly expanded tissue-resident T cell clones and the repertoire found in periphery blood samples. To trace and quantify donor reactive T cells the investigators will apply a truly quantitative approach for immune repertoire profiling based on high- throughput sequencing. The investigators ultimate goal is to develop a diagnostic tool to assess alloreactive cellular immunoresponses based on peripheral blood samples.

DETAILED DESCRIPTION:
Kidney transplant recipients receiving a non lymphodepletional induction therapy at the investigators center will be included in this study.

Alloreactive T cells are defined prior to transplantation via a mixed lymphocyte reaction of donor and recipient PBMC's.

Following transplantation PBMC's will be sampled at management (3 and 12 months) and for-cause biopsies and fifteen patients with histological proven acute T cell mediated rejection will be compared to 15 patients without histopathological signs of alloimmune response in time matched for-cause biopsies.

T cell receptor beta chains of T cells found in the circulation and the allograft biopsy will be sequenced via Next generation sequencing.

Abundance of alloreactive T cells of the overall repertoire pre-and post-transplant and their presence in the allograft will be assessed.

The diversity of the overall repertoire and alloreactive repertoire will be compared between these two groups.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplantation in our center

Exclusion Criteria:

* Donor not evaluated by our center

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Chronic kidney disease
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Rejection | 12 months
  biopsy proven rejection

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Oberbauer, MD, PhD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical university of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Aschauer C, Jelencsics K, Hu K, Heinzel A, Gregorich MG, Vetter J, Schaller S, Winkler SM, Weinberger J, Pimenov L, Gualdoni GA, Eder M, Kainz A, Troescher AR, Regele H, Reindl-Schwaighofer R, Wekerle T, Huppa JB, Sykes M, Oberbauer R. Prospective Tracking of Donor-Reactive T-Cell Clones in the Circulation and Rejecting Human Kidney Allografts. Front Immunol. 2021 Oct 14;12:750005. doi: 10.3389/fimmu.2021.750005. eCollection 2021. PMID 34721420
- [Derived] Aschauer C, Jelencsics K, Hu K, Heinzel A, Vetter J, Fraunhofer T, Schaller S, Winkler S, Pimenov L, Gualdoni GA, Eder M, Kainz A, Regele H, Reindl-Schwaighofer R, Oberbauer R. Next generation sequencing based assessment of the alloreactive T cell receptor repertoire in kidney transplant patients during rejection: a prospective cohort study. BMC Nephrol. 2019 Sep 2;20(1):346. doi: 10.1186/s12882-019-1541-5. PMID 31477052